CLINICAL TRIAL: NCT06835192
Title: Impact of Combining Course on Incontinence-associated Dermatitis Prevention and Management with Directive Wheel Chart for Nurses in Adult Wards
Brief Title: Impact of Combining Incontinence-associated Dermatitis Prevention and Management Course and Directive Wheel Chart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20240128
Record Dates: First submitted 2024-12-18; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Dermatitis; Knowledge, Attitudes, Practice
Keywords: Attitude; Course; Directive wheel chart; Incontinence-associated dermatitis; Knowledge; Practice
MeSH Terms: conditions — Dermatitis; Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: pretest-posttest design
Masking Description: educational intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Combining Incontinence-associated Dermatitis Prevention and Management Course and Directive Wheel Chart
  Interventions: Other: Experimental group; Other: Control Group
- Control Group (Other): The first author conducted a 25-minute knowledge lecture for the nurses in the CG on the same topics covered in the EG. This lecture included an explanation of IAD, its causes, the latest global classification of IAD, as well as methods for skin prevention and IAD care. Following the lecture, the same three clinical examples presented in the EG were discussed for an additional 20 minutes, during which the nurses were divided into groups for case discussions. Finally, a 5-minute quiz competition was held, featuring the same five actual clinical photographs used in the EG.
  Interventions: Other: Experimental group; Other: Control Group

INTERVENTIONS:
Other: Experimental group — Initially, the first author presented a 25-minute lecture with a PowerPoint presentation to the nurses of the EG. Following this, each nurse received an IAD directive wheel chart. In the subsequent 25 minutes, the first author presented three clinical cases examples and relevant information, encouraging the nurses to utilize the IAD directive wheel chart in groups. To conclude the session, a 5-minute quiz was conducted, featuring five actual clinical photographs. After the course, the nurses were instructed to take the IAD directive wheel chart back to their clinics for review and use in health education and teaching.
  Other Names: Combining Incontinence-associated Dermatitis Prevention and Management Course and Directive Wheel Chart
Other: Control Group — The first author conducted a 25-minute knowledge lecture for the nurses in the CG on the same topics covered in the EG. This lecture included an explanation of IAD, its causes, the latest global classification of IAD, as well as methods for skin prevention and IAD care. Following the lecture, the same three clinical examples presented in the EG were discussed for an additional 20 minutes, during which the nurses were divided into groups for case discussions. Finally, a 5-minute quiz competition was held, featuring the same five actual clinical photographs used in the EG.
  Other Names: Incontinence-associated Dermatitis Prevention and Management Course

SUMMARY:
Background: Knowledge, attitudes, and behaviors regarding the prevention and care of incontinence-associated dermatitis (IAD) need to be enhanced through educational training. There is a lack of innovative courses and convenient tools to assist nursing staff in learning and teaching in clinical settings.

Purpose: This study aims to investigate the learning outcomes of nursing staff in adult wards regarding the prevention and care of IAD, comparing the effectiveness of a course combined with an Directive Wheel Chart versus a course alone. Additionally, the study examines the effectiveness of nursing staff applying the course and Directive Wheel Chart in peer teaching.

DETAILED DESCRIPTION:
Design: This study was a two-phase randomized controlled trial conducted at a regional teaching hospital in Taiwan.

Materials and Methods: The study involved eight wards, comprising a total of 106 nurses, who were initially randomly assigned to either an experimental group (EG) or a control group (CG). Subsequently, the nurses within each ward were randomly allocated to two phases. The researcher delivered a 50-minute lecture to both groups, providing the IAD directive wheel chart only to the nurses in the EG. After a two-weeks period, one or two nurses from each ward in the first phase utilized the same course and directive wheel chart to peer-teach the nurses in the second phase within the same wards. The Chinese version of the Knowledge, Attitudes and Practices of Incontinence-associated Dermatitis Questionnaire (KAP-IAD-Q-C) and the Chinese version of the attitude towards the prevention of incontinence-associated dermatitis instrument (APrIAD-C) were employed to evaluate effectiveness. The Generalized Estimating Equation (GEE) was utilized to analyze the effectiveness of the educational intervention for each phase.

ELIGIBILITY:
Inclusion Criteria:

(1)Nurses in the eight adult wards.

Exclusion criteria:

1. New nurses had not completed the three-month probation period;
2. Nurses are holding administrative management positions
3. Nurse practitioners;
4. Nurses who expected to be employed within six months due to job transitions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The incontinence associated dermatitis knowledge, attitude and practice questionnaire (KAP-IAD-Q) | Four weeks prior to the course, after the teaching courses, four weeks after the course
  The total score ranges from 22 to 110 with higher scores indicating better the knowledge, attitude, and practical behaviors concerning IAD.
The attitude towards the prevention of incontinence-associated dermatitis instrument (APrIAD) | Four weeks prior to the course, after the teaching courses, four weeks after the course
  The questionnaire consists of 14 questions, each scored on a 4-point Likert scale., with a total score ranging from 0 to 42.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ting Su, BSN, Principal Investigator — Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung Medical University, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No